CLINICAL TRIAL: NCT07191301
Title: "Functional Strength Training and Kinesiotaping With and Without Proprioceptive Neuromuscular Facilitation Technique in Fibular (Peroneal) Neuropathy"
Brief Title: Functional Strength Training and Kinesiotaping, With and Without Proprioceptive Neuromuscular Facilitation in Fibular (Peroneal) Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Sumayyah Farooq, Sumayyah Farooq, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sumayah Farooq
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Peroneal Neuropathy
MeSH Terms: conditions — Peroneal Neuropathies | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group A (Experimental): Functional Strength Training (FST) + Kinesio Taping (KT) with Proprioceptive Neuromuscular Facilitation (PNF).
  Interventions: Behavioral: Functional Strength Training, Kinesio Taping, and Proprioceptive Neuromuscular Facilitation; Behavioral: Functional Strength Training and Kinesio Taping
- Control Group B (Active Comparator): Functional Strength Training (FST) + Kinesio Taping (KT) without PNF.
  Interventions: Behavioral: Functional Strength Training, Kinesio Taping, and Proprioceptive Neuromuscular Facilitation; Behavioral: Functional Strength Training and Kinesio Taping

INTERVENTIONS:
Behavioral: Functional Strength Training, Kinesio Taping, and Proprioceptive Neuromuscular Facilitation — Participants will undergo 8 weeks of supervised treatment, 3 sessions per week (24 sessions). Each session includes a warm-up with stretches, range-of-motion exercises, and Functional Strength Training (mini hops, stair climbing, ramp walking, sit-to-stand). Kinesio Taping will be applied from the foot's dorsum along the tibialis anterior and peroneus longus with 25-50% stretch for ankle support and dorsiflexor facilitation, re-applied every 3-4 days. In addition, Proprioceptive Neuromuscular Facilitation (PNF) lower-limb D1 flexion/extension patterns with manual resistance will be performed in 3 sets of 5 repetitions, lasting 35-40 minutes per session.
Behavioral: Functional Strength Training and Kinesio Taping — Participants will undergo 8 weeks of supervised treatment, 3 sessions per week (24 sessions). Each session includes a warm-up with stretches, range-of-motion exercises, and Functional Strength Training (mini hops, stair climbing, ramp walking, sit-to-stand). Kinesio Taping will be applied from the foot's dorsum along the tibialis anterior and peroneus longus with 25-50% stretch for ankle support and dorsiflexor facilitation, re-applied every 3-4 days. No PNF techniques will be applied.

SUMMARY:
Fibular neuropathy frequently manifests as foot drop, muscle weakness, altered gait, and sensory loss, all of which severely reduce mobility and quality of life. There is still uncertainty regarding the efficacy of kinesio taping (KT), proprioceptive neuromuscular facilitation (PNF), and functional strength training (FST) in combination. Although PNF improves neuromuscular coordination, KT provides proprioceptive input, and FST increases strength and mobility, there are no set treatment guidelines and little research has compared these modalities. In order to contribute to evidence-based rehabilitation techniques for people with fibular neuropathy, this study attempts to assess whether adding PNF to FST and KT improves functional outcomes compared to FST and KT alone.

ELIGIBILITY:
Inclusion Criteria:

* • Adults (18-35 years old) are diagnosed with fibular neuropathy due to trauma or compression.

  * Patients with muscle weakness, impaired balance and abnormal gait.
  * Both Male and female participants will be included.
  * Patients who test positive to the drag or slap test will be considered positive if the patient have difficulty in lifting the forefoot while walking, leading to dragging of the toes or compensatory hip/knee movements.

Exclusion Criteria:

* • Recent foot or ankle surgery (<6 months).

  * Complete loss of nerve supply
  * Severe musculoskeletal or neurological conditions (Amyotrophic lateral sclerosis, multiple sclerosis, myopathies, severe osteoarthritis, severe compression, progressive neuropathies, severe balance and fall risk, Guillain-Barré Syndrome (GBS) and peripheral vascular diseases).
  * Allergies to Kinesio tape materials.
  * Patients who are not psychologically fit such as those who have undergone trauma and patients with severe psychological disorders (major depressive disorder, PTSD, schizophrenia) will be excluded if they have had a diagnosis within the last 6 months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in dorsiflexor muscle strength measured by Manual Muscle Grading (MMG) | Baseline (Week 0), Mid-point (Week 4), and Post-intervention (Week 8)

IPD SHARING:
Plan to Share IPD: No